CLINICAL TRIAL: NCT01986140
Title: Scalp Cooling for Alopecia Prevention (SCALP)
Brief Title: Scalp Cooling to Prevent Chemo-induced Hair Loss
Acronym: SCALP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Julie Nangia (Other)
Responsible Party: Sponsor-Investigator, Julie Nangia, Assistant Professor, Baylor Breast Care Center
Organization: Baylor Breast Care Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H: 33692 SCALP
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Breast Cancer; Alopecia
Keywords: Breast Cancer; Alopecia; Scalp; Cooling
MeSH Terms: conditions — Breast Neoplasms; Alopecia

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: One blinded observer assesses the patient outcome
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PAXMAN Orbis Scalp Cooler (Experimental): Scalp Cooling
  Interventions: Device: PAXMAN Orbis Scalp Cooler
- Control No treatment (Other): Control
  Interventions: Other: Control No treatment

INTERVENTIONS:
Device: PAXMAN Orbis Scalp Cooler — Treatment with Orbis scalp cooling cap
  Arms: PAXMAN Orbis Scalp Cooler
Other: Control No treatment — No treatment to prevent hair loss
  Other Names: No intervention
  Arms: Control No treatment

SUMMARY:
Determine that the Orbis Paxman Hair Loss Prevention System is safe and effective in reducing chemotherapy-induced alopecia in woman with breast cancer undergoing neoadjuvant or adjuvant chemotherapy.

DETAILED DESCRIPTION:
Cooling the scalp during chemotherapy may help reduce the chances of losing hair during treatment. The investigators are hoping that using the PAXMAN Orbis Scalp Cooling Device may stop patients who are undergoing chemotherapy from losing their hair.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of breast cancer stage 1-2
* Planning to undergo neoadjuvant or adjuvant chemotherapy with curative intent
* Chemotherapy must be planned for at least 4 cycles of full-dose anthracycline or taxane based chemotherapy regimen,
* Defined as one of the following regimens: - Adriamycin 60mg/m2 with cyclophosphamide 600mg/m2 - Epirubicin 90-100mg/m2 with cyclophosphamide 600mg/m2 - Doxorubicin 50mg/m2 with 5-Fluroruacil 500mg/m2 and Cyclophosphamide 500mg/m2 - Paclitaxel 80mg-90/m2 weekly (every three weeks constitute a cycle), or 175 mg/m2 every 2-3 weeks as a single agent - Docetaxel 100mg/m2 as a single agent - Docetaxel 75mg/m2-100mg/m2 with pertuzumab and traztuzumab at standard doses - Docetaxel 75mg/m2 with cyclophosphamide 600mg/m2 - Docetaxel 75mg/m2 with carboplatin AUC of 6 and trastuzumab at standard doses
* Concurrent traztuzumab at standard doses is allowed
* Concurrent pertuzumab at standard doses is allowed
* Administration of chemotherapy on a dose dense schedule is allowed as clinically indicated.
* Subjects must have TSH collected within 1 year prior to treatment and found within normal range.
* If patient has a history of diabetes, Hemoglobin A1c must be drawn within 3 months prior to treatment and found to be within normal limits.
* CBC and CMP should be done within 4 weeks prior to treatment and found to be within acceptable limits.

Exclusion Criteria:

* Stage 3 or 4 breast cancer or any other concurrent malignancy including hematological malignancies (i.e. leukemia or lymphoma)
* Baseline alopecia (defined CTCAE v4.0 grade > 0, see appendix B for CTCAE v4.0 scale)
* Subjects with cold agglutinin disease or cold urticaria
* Subjects who are scheduled for bone marrow ablation chemotherapy
* Subjects receiving chemotherapy with concurrent anthracycline and taxane (AT or TAC)
* Male gender
* Age >= 70 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2014-05-15 (Actual); Primary Completion 2017-02-10 (Actual); Study Completion 2022-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Nangia, M.D., Principal Investigator — Baylor College of Medicine
Locations (7):
- United States (7):
  - Hematology & Oncology Associates of Northern New Jersey, Morristown, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Texas Oncology - Medical City Dallas, Dallas, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - USOncology / Texas Oncology-Memorial City, Houston, Texas
  - Lester and Sue Smith Breast Center at Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Patients are aware of whether or not they are using the cooling device and can tell if they have hair loss.
Supporting Information: ICF
Time Frame: At completion of their participation.
Access Criteria: Patients know if they are wearing the device or not.

REFERENCES:
- [Derived] Chevli N, Wang K, Haque W, Schwartz MR, Nangia J, Sasaki J, Farach AM, Hatch SS, Butler EB, Teh BS. Prognostic Impact of Radiation Therapy in Pure Mucinous Breast Carcinoma. Clin Breast Cancer. 2022 Oct;22(7):e807-e817. doi: 10.1016/j.clbc.2022.06.005. Epub 2022 Jul 7. PMID 35915020
- [Derived] Nangia J, Wang T, Osborne C, Niravath P, Otte K, Papish S, Holmes F, Abraham J, Lacouture M, Courtright J, Paxman R, Rude M, Hilsenbeck S, Osborne CK, Rimawi M. Effect of a Scalp Cooling Device on Alopecia in Women Undergoing Chemotherapy for Breast Cancer: The SCALP Randomized Clinical Trial. JAMA. 2017 Feb 14;317(6):596-605. doi: 10.1001/jama.2016.20939. PMID 28196254

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PAXMAN Orbis Scalp Cooler | Control No Treatment
Started (subjects who were randomized) | 157 | 79
Completed (subjects who underwent scalp cooling or non-cooling for a 4 cycles of chemotherapy) | 122 | 51
Not Completed | 35 | 28
Not completed — Withdrawal by Subject | 31 | 25
Not completed — alternative treatment | 1 | 1
Not completed — found not eligible | 3 | 0
Not completed — Adverse Event | 0 | 1
Not completed — progression disease | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Scalp Cooling: Scalp Cooling
  PAXMAN Orbis Scalp Cooler: Treatment with Orbis scalp cooling cap
- Non-cooling: Control
  Control No treatment: No treatment to prevent hair loss
- Total: Total of all reporting groups
Arm/Group | Scalp Cooling | Non-cooling | Total
Number analyzed (Participants) | 157 | 79 | 236
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (10.1) | 50.6 (10.6) | 50.4 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 157 | 79 | 236
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 12 | 37
  Not Hispanic or Latino | 130 | 66 | 196
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 10 | 29
  White | 130 | 62 | 192
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 157 | 79 | 236

OUTCOME MEASURES:

1. Primary Outcome: Hair Preservation
Description: The primary efficacy endpoint will be success in hair preservation, defined as CTCAE v 4 alopecia grade <2, and will be assessed by a healthcare professional who is blinded to study treatment.
Time Frame: 4 to 8 Months
Population: Randomized patients who underwent at least one cycle of chemotherapy were evaluable for efficacy. 27 patients in the cooling group and 25 patients in the non-cooling group did not start chemotherapy or discontinued during the 1st cycle were excluded from the efficacy analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Scalp Cooling | Non-cooling
Number analyzed (Participants) | 130 | 54
Participants
  success | 69 | 0
  failure | 61 | 54

2. Secondary Outcome: Time to First Recurrence and Overall Survival
Description: A safety follow-up for safety data will be done yearly for 5 years looking at time to first recurrence of breast cancer, overall survival, site of first recurrence, and incidence of isolated scalp metastasis. This will be collected during routine clinical observation
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2022-02

3. Other Pre Specified Outcome: Improved Quality of Life
Description: Improved quality of life as a result of reduced hair loss is a primary motivator for developing the Paxman Scalp Cooling device. Quality of life will be assessed at baseline and 2-3 weeks after each course of chemotherapy. Three widely used and validated scales will be used: the EORTC QLQ C-30, HADS and BIS. Subjects will be evaluated at multiple time points and data will be analyzed using descriptive methods with median and inter quartile rang to assess the effect of treatment group and alopecia status on functioning, quality of life and depression.
Time Frame: 4 to 8 Months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events experienced by subjects were collected from initiation of study device, throughout the study for up to 8 cycle of device use, and within 30 days of the last use of study device. Adverse events through 30 days after study completion were collected.
Description: Any adverse events that are possibly, probably, or definitely related to the Orbis Paxman Hair Loss Prevention System were reported. Any toxicities were determined to be related to the chemotherapy were monitored and only reported if they were unusual. Subjects who were randomized to the scalp cooling and started the first cycle of chemotherapy were evaluable for safety analyses.
  No adverse event from non-cooling subjects since they did not use the device so they were not at risk.
Arm/Group | Scalp Cooling | Non-cooling
All-Cause Mortality (participants affected / at risk) | 0/137 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/137 | 0/0
Other Adverse Events (participants affected / at risk) | 39/137 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Scalp Cooling (N=137) | Non-cooling (N=0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 7 (11) | 0 (0)
chills (General disorders) | 1 (1) | 0 (0)
pain (General disorders) | 1 (1) | 0 (0)
dizziness (Nervous system disorders) | 6 (7) | 0 (0)
headache (Nervous system disorders) | 27 (34) | 0 (0)
paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Sinus pain (Nervous system disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
scalp pain (Skin and subcutaneous tissue disorders) | 6 (7) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-07-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT01986140/Prot_000.pdf
  • Statistical Analysis Plan (2015-11-30): https://cdn.clinicaltrials.gov/large-docs/40/NCT01986140/SAP_003.pdf
  • Informed Consent Form (2016-07-06): https://cdn.clinicaltrials.gov/large-docs/40/NCT01986140/ICF_001.pdf